CLINICAL TRIAL: NCT04384783
Title: To Explore the Effect of Low-dose Long Term Growth Hormone Pretreatment on Clinical Pregnancy Outcomes in Patients With Low Ovarian Reserve
Brief Title: To Explore the Effect of GH Pretreatment on Clinical Outcomes in Patients With Low Ovarian Reserve
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20201A011002
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: GH; Low Ovarian Reserve
Keywords: GH; low ovarian reserve; POSEIDON
MeSH Terms: interventions — Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GH group: GH group: Participants diagnosed POR according to POSEIDON criteria with low ovarian reserve undergo IVF in our center with long protocol or antagonist protocol and is adjuvant with GH 2IU/d from previous menstrual period for about six weeks.
  Interventions: Drug: growth hormone
- NGH group: NGH (non-GH) group: Participants diagnosed POR according to POSEIDON criteria with low reserve undergo IVF in our center with long protocol or antagonist protocol without GH adjuvant.

INTERVENTIONS:
Drug: growth hormone — growth hormone was adjuvanted 2IU/d from previous menstrual period for about six weeks.
  Groups: GH group

SUMMARY:
Growth hormone (GH) has been used in the field of assisted reproduction technology for over 30 years. Studies for GH have been exploring in the applicable population, drug dosage, starting time and time limitation. In previous clinical applications, it worked as an adjuvant drug for improving ovarian reactivity. With the development of basic research and clinical applications, the improvement effect on egg quality is gradually recognized. However, which protocol of GH may work well and maximize the clinical effect remains mystery. The investigators' previous self-controlled retrospective research about 380 cases treated with GH found that the average daily injection of GH dose of 2IU for about 6 weeks can significantly improve embryo quality and clinical pregnancy outcomes of the patients with low ovarian response. The new POSEIDON standard clearly groups people with low prognosis and better classifies heterogeneous people, which may help classifying the specific subgroup that benefit most from GH of poor ovarian response (POR). The investigators design a prospective cohort study to explore whether GH low-dose long-term pretreatment can improve the outcome of assisted pregnancy and its possible mechanism in people with low ovarian reserve.

ELIGIBILITY:
Inclusion Criteria:

1. low ovarian reserve(AMH <1.2ng/ml, or AFC <5);
2. patients who have not participated in any clinical trials within the three months;
3. patients who voluntarily signed informed consent.

Exclusion Criteria:

1. patients with BMI ≥30kg/m2;
2. patients with medical diseases such as endocrine and metabolic diseases, autoimmune disease, etc;
3. ovarian neoplasm that ≥4 cm in diameter and has no clear pathological diagnosis by surgery;
4. complicated with adenomyosis, endometriosis confirmed by surgery;
5. patients with untreated abnormal intrauterine environment, such as uterine effusion, endometritis, etc;
6. untreated hydrosalpinx.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients enroll for study are based on POSEIDON criteria[1], and with informed consent.
Sampling Method: Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2020-05-26 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
rate of good quality embryos | 2 years
  the number of good quality embryos divide by the number of transferrable embryos

SECONDARY OUTCOMES:
number of oocytes retrieved | 2 years
  number of oocytes retrieved
fertilization rate | 2 years
  the fertilized oocytes divided by the number of oocytes retrieved
clinical pregnancy rate | 2 years
  the patients confirmed clinical pregnancy divided by the patients undergoing fresh embryo transferred.
live birth rate | 2 years
  the patients have a live birth divided by the patients undergoing fresh embryo transferred.

CONTACTS AND LOCATIONS:
Overall Officials: meihong Cai, master, Study Director — Guangzhou First People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Poseidon Group (Patient-Oriented Strategies Encompassing IndividualizeD Oocyte Number); Alviggi C, Andersen CY, Buehler K, Conforti A, De Placido G, Esteves SC, Fischer R, Galliano D, Polyzos NP, Sunkara SK, Ubaldi FM, Humaidan P. A new more detailed stratification of low responders to ovarian stimulation: from a poor ovarian response to a low prognosis concept. Fertil Steril. 2016 Jun;105(6):1452-3. doi: 10.1016/j.fertnstert.2016.02.005. Epub 2016 Feb 26. No abstract available. PMID 26921622